CLINICAL TRIAL: NCT03533400
Title: The Effectiveness of the Jamboxx Respiratory Therapy Device in Treatment of Patients With Decreased Respiratory Function. Study 1: Spinal Cord Injury Patients for Long Term Evaluation
Brief Title: Effectiveness of Jamboxx Respiratory Therapy Device: Study 1
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: NHLBI has suggested the company focus on the other two ongoing trials
Sponsor: My Music Machines Inc. (Industry)
Collaborators: Albany Medical College (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Jamboxx RT Device Study 1; 4R42HL132735-02 (NIH)
Record Dates: First submitted 2018-04-26; First posted 2018-05-23 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Spinal Cord Injuries; Respiratory Complication
Keywords: respiratory therapy; videogaming therapy; incentive spirometry
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: Study participants will be randomized into 2 groups via random number generator. Group 1 (control group) will be given the standard Jamboxx musical device, while Group 2 (treatment group) will be given the Jamboxx respiratory therapy device, which combines musical gameplay with incentive spirometry exercises.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Group 1 (Active Comparator): Group 1 (control group) will be given the standard Jamboxx musical device. They will be trained to use the device during two 20 minute training session with a respiratory therapist, and will be instructed to play the device for a minimum of 30 minutes, 3 times a week. The Jamboxx musical device is a hands-free breath controlled musical device designed for people with quadriplegia. The mouthpiece acts as a transducer, changing air pressure created by the user's lungs to a joystick signal to the computer via a differential pressure sensor. The Jamboxx can produce musical sounds of many instruments (trumpet, drums, etc.) in many different scales and in any key.
  Interventions: Device: Jamboxx Musical Device
- Group 2 (Experimental): Group 2 (treatment group) will be given the Jamboxx musical device plus the Jamboxx respiratory therapy device. The respiratory therapy device is similar to the music device, but with specially designed games that guide the user through breathing exercises intended to strengthen the lungs.
  Interventions: Device: Jamboxx Respiratory Therapy Device; Device: Jamboxx Musical Device

INTERVENTIONS:
Device: Jamboxx Respiratory Therapy Device — Jamboxx Respiratory Therapy Device is a novel device that uses interactive gaming to encourage patient compliance with their prescribed respiratory therapy routines. The device consists of a computer game controller with mouthpiece containing a breath flow sensor that connects to a tablet. With the Jamboxx respiratory therapy device, users can choose from a suite of breath controlled respiratory therapy games to guide them through their routines while receiving real-time feedback, and long-term progress tracking.
  Arms: Group 2
Device: Jamboxx Musical Device — Jamboxx musical device is a hands free, breath controlled music device designed for people with quadriplegia. It resembles a common harmonica in that the user slides a mouthpiece along its horizontal axis to change the pitch of the instrument. The device connects to a personal computer via a mini USB to USB cable to interface with software that provides visual feedback for playing notes and sends the information to the computer speakers. The mouthpiece acts as a transducer, changing air pressure created by the user's lungs to a joystick signal to the computer via a differential pressure sensor. The Jamboxx musical device can produce musical sounds of many instruments (trumpet, drums, etc.) in many different scales and in any key

SUMMARY:
The Effectiveness of the Jamboxx Respiratory Therapy Device in Treatment of Patients with Decreased Respiratory Function is a proposal for investigation of the application of gaming to improving respiratory health. The Jamboxx device combines gaming with traditional incentive spirometry to provide users with a fun experience to keep them engaged in their respiratory therapy routine. The device allows users to play a series of mini-games that walk them through their routines. The Jamboxx also records airflow and lung parameters with an external mouthpiece attachment to provide users with real time feedback, and helps to assess increases or decreases in relative lung function over time. The Jamboxx has the potential to significantly impact the field of respiratory therapy by being one of the first gaming devices for patient therapy, and the first respiratory therapy gaming device that is accessible to users with limited mobility. Jamboxx provides a fun and engaging, low cost alternative to the traditional therapy techniques used and aims to improve patient compliance.

DETAILED DESCRIPTION:
Study 1 addresses the concerns of pneumonia risks in quadriplegics with compromised respiratory pump mechanics. In cases of spinal cord injury or high-level motor neuron disease, complications with respiratory function are a common concern. Lack of innervation to the intercostal and abdominal muscles can cause a decline in respiratory capacity as well as overall lung function, with associated increased risk of mortality. Shallow tidal breathing and impaired or absent cough results in morbidity and mortality from pneumonia. Several studies have found failure of the respiratory system, including pneumonia, to be a leading cause of mortality among spinal cord injury patients. In order to maintain pulmonary health, many people with quadriplegia and other high-level motor neuron diseases undergo routine respiratory therapy to help stretch the muscles around the lungs, exercise the diaphragm, and loosen mucus build-up. Incentive spirometry is one commonly used component of respiratory therapy designed to mimic natural sighing or yawning by encouraging the patient to take long, slow, deep breaths. This is done with an incentive spirometer device, which provides patients with visual or other positive feedback with a piston or a ball that moves inside a gauge. Respiratory therapy techniques are also used to help maintain pulmonary health in individuals with a number of chronic or temporary respiratory diseases and conditions such as asthma, chronic obstructive pulmonary disease, and emphysema. These techniques often become strenuous and mundane for users with limited mobility, and thus patient compliance rates are low. Gaming controlled by forceful respiratory maneuvers will be studied to ascertain if respiratory mechanics can be improved in this group.

Testing Plan: Study participants will be randomized into 2 groups through drawing of sealed envelopes. Group 1 (control group) will be given the standard Jamboxx musical device (see appendix a for device details), while Group 2 (treatment group) will be given the Jamboxx respiratory therapy device, which combines musical gameplay with incentive spirometry exercises. Participants from both groups will have two 20 minute training sessions with the device: one initial training visit and one follow up visit. Training sessions will take place either in the home, or at Albany Medical Center. During the initial visit a simple spirometry test (FEV1, FVC and PEF) and maximum inspiratory and expiratory pressures (MIP and MEP) will be performed. These functions will be measured again at 3, 6, 9 & 12 months by a respiratory therapist (RT). The Dyspnea-12 (D-12) questionnaire will be conducted at by the RT at months 0, 3, 6, 9, and 12. Self-Reported Patient Dyspnea and the Multidimensional Dyspnea Profile (MDP) will be reported electronically by study participants on a weekly basis. Medical records will be evaluated for relevant health history, medication use, and hospitalizations including dates. Access to medical records will be obtained by a signed medical release form.

ELIGIBILITY:
Inclusion Criteria:

* Quadriplegic and other spinal cord injury outpatients will be included.

Exclusion Criteria:

* Individuals already adhering to a daily regimen of prescribed respiratory therapy routine will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-12-01 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Self-Reported Patient Dyspnea | reported 1x/ week for the duration of the 1 year study
  Change in patient reported measure of breathlessness during daily activities from baseline over the course of the 1 year study

SECONDARY OUTCOMES:
Multidimensional Dyspnea Profile | reported 1x/ week for the duration of the 1 year study
  A measure of breathlessness after performing an activity
Dyspnea-12 Questionnaire | Months 0, 3, 6, 9, 12
  A survey that measures recent breathlessness with 12 questions related to dyspnea, each evaluated on a scale of 0-4 (0=none, 1=mild, 2=moderate, 3=severe) that indicate how troubled people are by each of these 12 topics, for a total possible score ranging from 0 to 36, where lower scores relate to better outcomes.
FEV1 | Months 0, 3, 6, 9, 12
  measure of pulmonary function (Forced Expiratory Volume over 1 second) measured in liters
FVC | Months 0, 3, 6, 9, 12
  measure of pulmonary function (Forced Vital Capacity) measured in liters
PEF | Months 0, 3, 6, 9, 12
  measure of pulmonary function (Peak Expiratory Flow) measured in liters
MEP | Months 0, 3, 6, 9, 12
  measure of pulmonary function (Maximum Expiratory Pressure) measured in centimeters of H2O
MIP | Months 0, 3, 6, 9, 12
  measure of pulmonary function (maximum inspiratory pressure) measured in centimeters of H2O
Device usability | Months 6, 12
  Measurement of enjoyment and engagement with the intervention via survey
Clinically relevant events | Months 0, 3, 6, 9, 12
  e.g. patient being sent for a chest x-ray, being ordered chest physiotherapy or blood tests
Patient Empowerment | Months 0, 3, 6, 9, 12
  Measured via a single question ranked on a likert scale: "I believe that this respiratory therapy empowered me to protect my breathing" With answer options of 1. strongly disagree, 2. disagree, 3. neutral, 4. agree, 5. strongly agree, with higher numbers corresponding to better outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Marilyn Fisher, MD, Study Chair — Albany Medical College
Locations (1):
- Albany Medical Center, Albany, New York, United States

IPD SHARING:
Plan to Share IPD: No